CLINICAL TRIAL: NCT00322504
Title: Acupuncture for Anxiety in Women With Breast Cancer: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0520C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2006-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Accupuncture

SUMMARY:
To assess the efficacy of acupuncture treatment in reducing symptoms of anxiety in women recently diagnosed with cancer.

• To assess the efficacy of acupuncture treatment on improving perceived quality of life in women recently diagnosed with cancer.

DETAILED DESCRIPTION:
This is a feasibility study of acupuncture for anxiety reduction in women with breast cancer. Ten patients will be recruited at the UNM Cancer Research Treatment Center via the Breast Clinic and screened for anxiety. Treatment will consist of 10 acupuncture sessions over 5 weeks. Measures (Hopkins Symptom Checklist, Sheehan Disability Index) will be administered and analyzed for treatment effect on scores.

ELIGIBILITY:
Inclusion Criteria:

* Woman age 18 years or older excluding the need for parental/guardian permission.
* Histologic diagnosis of breast cancer.
* Having a minimum anxiety score of 1.75 on the Hopkins Symptom Checklist (HSCL) with sufficient English language proficiency for the investigators to make this determination.
* Able to give informed consent.
* Willingness to participate in the study and receive 10 acupuncture treatments in 5 weeks.
* Ability to fill out questionnaires and communicate with the research staff

Exclusion Criteria:

* Males with breast cancer
* Psychoses or a major personality disorder
* Current use of opiates,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-01; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shelley, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States